CLINICAL TRIAL: NCT05767684
Title: Personalized Neoantigen Derived Dendritic Cell-Based Immunotherapy as Cancer Treatment
Brief Title: Neoantigen Derived DCs as Cancer Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-108-087
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-02

CONDITIONS: Refractory Tumor; Solid Tumor
Keywords: immunotherapy; cancer vaccine; neoantigen
MeSH Terms: conditions — Neoplasms | interventions — lenvatinib; Nivolumab

STUDY DESIGN:
Intervention Model Description: All patient will receive DCs monotherapy initially on day 1, 8, 15 and 29 as safety run-in. Safety and efficacy (1st CT evaluation) will be conducted at day 43. On the 1st CT evaluation, patient met randomization criteria and without progression disease/safety concern will be randomized to either observation or booster of lenvatinib and nivolumab during day 43 to 77.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: DCs monotherapy (Experimental): DCs injection on day 1, 8, 15, 29, 85, 141, 197, 253 and 309.
  Interventions: Biological: Dendritic Cell Vaccine
- Arm 2: DCs with booster of anti-VEGF/anti-PD-1. (Experimental): DCs injection on day 1, 8, 15, 29, 85, 141, 197, 253 and 309 plus lenvatinib 10mg QD on day 43-77 and nivolumab 3mg/kg on day 43, 57 and 71.
  Interventions: Biological: Dendritic Cell Vaccine; Drug: Lenvatinib; Drug: Nivolumab

INTERVENTIONS:
Biological: Dendritic Cell Vaccine — Approximately 1.5 x 10^6±20% cells will be subcutaneously injected to the patient's inguinal area (either left side or right side can be injected, only one area will be injected each time) on day 1, 8, 15, 29, 85, 141, 197, 253 and 309.
  Other Names: DCs
Drug: Lenvatinib — Lenvatinib 10mg/day on day 43-77
  Other Names: Lenvima
  Arms: Arm 2: DCs with booster of anti-VEGF/anti-PD-1.
Drug: Nivolumab — Nivolumab 3mg/kg on day 43, 57 and 71.
  Other Names: OPDIVO
  Arms: Arm 2: DCs with booster of anti-VEGF/anti-PD-1.

SUMMARY:
Tumor lysate or carcinoembryonic antigen (CEA) derived DCs-based therapy is safe and can elicites remarkable T-cell responses but mostly did not really transfer into significant clinical benefit. One possible reason is the lack of effective antigen and the immunosuppressive microenvironment. Now we are exploring another new strategy, prediction of neoantigen for priming DCs as cell-based therapy with or without booster of anti-VEGF/anti-PD-1.

DETAILED DESCRIPTION:
The human immune system can recognize and destroy cancer cells but cancer cells are capable of escaping from immune system by different ways, including the PD-1/PDL-1 axis and the VEGF signaling pathway. The PD-1/PD-L1 axis represents an adaptive immune resistance mechanism exerted by tumor cells. Previous study also revealed VEGF-A could induce tumor-associated macrophages, Treg cells, and myeloid-derived suppressor cells, creating an immunosuppressive microenvironment that prevent the maturation of dendritic cells (DCs) and inhibit the activation of NK cells and T cells. Our research group already completed some early phase clinical trials of DCs-based therapy, which illustrated tumor lysate or carcinoembryonic antigen (CEA) derived DCs-based therapy is feasible and safe in patients with advanced colorectal cancer and lung cancer, respectively. However, although DCs-based therapy elicited remarkable T-cell responses but mostly did not really transfer into significant clinical benefit in previous study. One possible reason is the lack of effective antigen and the immunosuppressive microenvironment. Now we are exploring another new strategy, prediction of neoantigen for priming DCs as cell-based therapy with or without booster of anti-VEGF/anti-PD-1.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years of age
* Provide written informed consent
* Histologically confirmed stage IV pancreatic cancer, liver cancer, biliary tract cancer and colorectal cancer (excluding sarcoma and neuroendocrine tumor) that refractory or intolerance to standard therapies for their condition (there is no effective treatment by investigator judgement)
* Completed tumor and germline DNA and RNA sequencing and the neoantigen prediction
* Patients with chronic hepatitis B is eligible if receiving anti-hepatitis B agents and the HBV DNA level < 2000 IU/ml prior to the preparation phase. Patients with chronic hepatitis C are eligible if HCV RNA is undetectable (<15 IU/ml) prior to the preparation phase
* Adequate organ function

  * Absolute neutrophil count >1000/mcL
  * Hemoglobin > 8.0 g/dl
  * Platelet > 50000/mcL
  * PT/aPTT < 1.5 x upper limit of normal (ULN)
  * AST/ALT < 3 x ULN
  * Bil(T) < 1.5 x ULN
  * BUN/Cr < 1.5 x ULN
* Adequate immune system as defined by

  * IgG > 614 mg/dl
  * IgM > 53mg/dl
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Life expectancy at least>12weeks
* At least one measurable target lesion as defined by RECIST 1.1

Exclusion Criteria:

* Sarcoma、neuroendocrine tumor
* Last anticancer therapy administered within 2 weeks and any AEs should be ≤ grade 2 prior to leukapheresis
* Patients who cannot tolerate leukapheresis and follow-up blood sampling of 50ml at day 43, day 85 and end-of- treatment.
* Any known active infection as judged by the investigator
* Any known chronic active infection of HIV, HTLV-1 or HTLV-2
* Requirement of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to the screen phase. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Other immunocompromising condition that in the opinion of the treating physician renders the patient a poor candidate for this trial
* Pregnant women, nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device (IUD), abstinence, etc.)
* Patients with history of penicillin allergy
* Other medical problems or conditions that, in the opinion of the investigator, would make participation in the study hazardous for the patient

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experienced limiting toxicities in the first 6 weeks. | 6 weeks
  The following toxicities that happened during first 6 weeks are considered LTs. Toxicities are graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0:
  * >=Grade 3 non-hematological toxicity
  * >=Grade 4 hematological toxicity
  * Any death not clearly due to the underlying disease or extraneous causes.
  * Any case meeting Hy's law
  * Recurrent grade 2 pneumonitis

SECONDARY OUTCOMES:
Percentage of patients who had a clinical response | 1 year
  Response was assessed by the iRECIST.
Number of participants who did not progressed or survived at 1 year | 1 year
  1 year progression-free survival and overall survival rate
Number of subjects experienced any ≥ grade 3 toxicities. | 1 year
  any ≥ grade 3 toxicities rate

OTHER OUTCOMES:
Number of subjects experienced immune response | 1 year
  The production of IFN-γ that occurs subsequent to the dendritic cells-based therapy as determined by ELISPOT Assay or Flow Cytometry Analysis. Other immune response biomarker study including but not limited to whole exome sequencing, bulk RNA sequencing and single cell RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, MD, PhD, Principal Investigator — Kaohsiung Medical University Hospital, and Center for Cancer Research, Kaohsiung Medical University
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Cheng-Kung University Hospital, Tainan
  - National Institute of Cancer Research, Tainan

IPD SHARING:
Plan to Share IPD: No